CLINICAL TRIAL: NCT01472276
Title: Effect of a Unique Web-based Behaviour Change Program for Physical Activity and Weight Management on Weight Loss and Cardiovascular Risk Factors in Overweight or Obese Adults at High Risk of Cardiovascular Disease
Brief Title: Effect of a Unique Web-based Behaviour Change Program on Weight Loss and Cardiovascular Risk Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: AXA PPP Healthcare (Industry)
Responsible Party: Principal Investigator, Michelle McKinley, Lecturer, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10041MMcK-OPMS; 10/NIR02/28 (Other: ORECNI)
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-06

CONDITIONS: Obesity
Keywords: Behaviour change; Weight loss; Cardiovascular risk; Diet; Physical activity; Overweight; Obesity; Internet
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Web-based program (Active Comparator)
  Interventions: Behavioral: Web-based program

INTERVENTIONS:
Behavioral: Web-based program — Provided with the web-based program
  Arms: Web-based program

SUMMARY:
Web- or internet-based programs have the potential to induce and, possibly, help to sustain, significant lifestyle modification. This study will evaluate the effect of a unique interactive web-based behaviour change program on weight loss and cardiovascular risk factors in people who are overweight or obese and at high risk of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Have regular access to the internet, telephone and have an e-mail address.
* Body mass index (BMI) greater than 27 and less than 40
* Sedentary
* Have one or more of the following risk factors associated with cardiovascular disease: Elevated blood pressure ≥ 140 mm Hg systolic or ≥ 90 mm Hg diastolic; Elevated total cholesterol ≥ 5.0; Type 2 diabetes
* Be willing to refrain from participating in another behaviour change program for the duration of the study

Exclusion Criteria:

* Major health problems including Type 1 diabetes, established CVD, renal and hepatic disease
* Psychiatric problems
* Pregnancy
* Excessive alcohol consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McKinley, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, Antrim, United Kingdom

REFERENCES:
- [Derived] Watson S, Woodside JV, Ware LJ, Hunter SJ, McGrath A, Cardwell CR, Appleton KM, Young IS, McKinley MC. Effect of a Web-Based Behavior Change Program on Weight Loss and Cardiovascular Risk Factors in Overweight and Obese Adults at High Risk of Developing Cardiovascular Disease: Randomized Controlled Trial. J Med Internet Res. 2015 Jul 16;17(7):e177. doi: 10.2196/jmir.3828. PMID 26183659

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Web-based Program
Started (Randomized) | 33 | 32
3-month Follow-up | 32 | 25
6-month Follow-up | 31 | 21
Completed (12-month follow-up) | 29 | 17
Not Completed | 4 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Web-based Program | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (7.27) | 51.4 (7.59) | 52.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss Kg
Description: Between-group change in weight loss at 3-month follow-up
Time Frame: 3 months
Population: Weight (kg) outcome differences within study groups from baseline to 3 months (complete-case analysis).
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Control | Web-based Program
Number analyzed (Participants) | 32 | 25
kg | -0.53 [-1.60 to 0.54] | -4.37 [-5.80 to -2.94]

2. Secondary Outcome: Weight Loss
Description: Between-group change in weight loss at 6 and 12 months
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Physical Activity
Description: Assessed by triaxial accelerometer and RPAQ questionnaire
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Blood Pressure (Seated, Systolic and Diastolic mmHg)
Description: Seated, systolic and diastolic mmHg
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Biochemical Markers of CVD Risk
Description: Total cholesterol HDL cholesterol, LDL cholesterol, triglycerides high-sensitivity CRP, HOMA, HbA1c
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Dietary Intake
Description: Diet history
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Pulse Wave Analysis
Description: SpygmoCor Pulse Wave Analysis System
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Quality of Life
Description: Questionnaire
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Sleep Quality
Description: Questionnaire
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Self-esteem
Description: Questionnaire
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

11. Secondary Outcome: Self-efficacy
Description: Questionnaire
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

12. Secondary Outcome: Depression
Description: Questionnaire
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control | Web-based Program
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes